CLINICAL TRIAL: NCT02914002
Title: A Psychoeducational Intervention Model in Nutrition to Improve Nutritional Status in 15 Low Resource Populations Through a Network of Food Banks in Mexico.
Brief Title: Psychoeducational Intervention Model to Improve Nutritional Status in Low Resource Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Monterrey (Other)
Collaborators: FEMSA Foundation (Other); Mexican Food Banks (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 502016-CIE
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Child Malnutrition; Child Overnutrition; Malnutrition in Children; Malnutrition, Child; Nutrition Disorders, Child; Malnutrition
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Psychoeducational intervention (Experimental): Participants will be receiving a cooking lesson in their community every 2 weeks for 1 year.
  Interventions: Behavioral: Psychoeducational intervention
- Usual Food Practices - AC (No Intervention): These are participants from the communities where the intervention is active but are not attending the cooking lessons.
- Usual Food Practices - NAC (No Intervention): These are participants from a community where the intervention is not active.

INTERVENTIONS:
Behavioral: Psychoeducational intervention — A mobile kitchen visits the 16 selected communities every 2 weeks for a period of 1 year. A 30 minute cooking lesson is given by a trained instructor, the recipes have been designed to be quick and easy to make, use local and inexpensive ingredients, contain mostly vegetables and have a good taste. During the lesson, healthy habit and cooking tips are mentioned as well as the importance of cooking at home and having family meals . A printed version of the recipe is given to every participant. Every session participants are encouraged to prepare the recipe. At the end of the lesson all the participants get to taste the meal and express their opinion.
  Other Names: Psychoeducational intervention in nutrition
  Arms: Psychoeducational intervention

SUMMARY:
Comer en Familia is a psychoeducational intervention in nutrition aimed to improve nutritional status in families, particularly mothers and caregivers of children between the ages of 5 and 13 years and their children through providing healthy cooking lessons in their communities where the optimal preparation and use of local foods based on vegetables is promoted at the same time the importance of cooking at home and eating as a family is highlighted.

DETAILED DESCRIPTION:
It is well known that in order to promote a proper nutrition and to prevent malnutrition in Mexican population, both by deficiencies and excesses, it is essential to recover Mexican food culture. It is known that only information is insufficient to implement healthy lifestyles. There are a number of barriers that interfere with the adoption of healthy dietary practices that need to be identified and addressed in order to achieve the adoption of healthy eating behaviors. Therefore, Comer en Familia focuses on the people, their lifestyles, motivations and social context, based on an action methodology. To design the program, culinary traditions from different country regions were integrated, the habits of proper food preparation at home, promoting eating in the company of family with special emphasis on the importance of enjoying the taste of food were also integrated. This model delivers information on the transcendence of preparing food at home, the impact of nutrients on health and the influence of eating habits of the family in the conducts of their members in a practical way. Comer en Familia is a nutritional educational model that aims to promote proper nutrition, and therefore improve health and welfare of the beneficiaries of food banks. Through 24 cooking workshops throughout a period of a year, each workshop every 15 days, communities will be trained in optimal food preparation and the use of local food, based mainly on vegetables, while promoting the importance of cooking and having family meals. Anthropometric evaluations and interviews on food practices will be conducted to the beneficiaries at the beginning and at the end of the program. Anthropometric evaluations will be carried out and psychosocial risks surveys will be applied to the children in charge of the mothers/ caregivers from Comer en Familia. Also, in a sub-sample of the population of mothers/caregivers benefitted from the program, fasting capillary glucose and hemoglobin will be measured at the beginning and at the end of Comer en Familia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years
* Premenopausal
* Related to the decision of purchase, planning, elaboration-preparation of meals at home.
* Not being pregnant during the period of the study or the six prior months, and planning not to be pregnant at least 3 months after the last visit of the study.
* With a child in her care between the ages of 5 and 13 years and that fulfills the inclusion criteria

Exclusion Criteria:

* Pregnant or breastfeeding
* With a hysterectomy in the past 3 months
* Alcohol consumption > 14 drinks a week
* Use of vitamin supplements

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12400 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Change in food knowledge and behavior Questionnaire | Baseline, 1 year
Change in Weight | Baseline, 1 year
Change in height | Baseline, 1 year
Change in psychosocial risk Questionnaire | Baseline, 1 year

SECONDARY OUTCOMES:
Change in capillary hemoglobin | Baseline, 1 year
  Capillary blood sample
Change in capillary glucose | Baseline, 1 year
  Capillary blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Ana Carla Cepeda-Lopez, PhD, Principal Investigator — Universidad de Monterrey
Locations (1):
- Banco de Alimentos de Mexico, México, Mexico

IPD SHARING:
Plan to Share IPD: No